CLINICAL TRIAL: NCT00931190
Title: Evaluation of the Use of Human Papillomavirus Persistence for Determination of the Treatment Efficacy Among Women With Cervical Intraepithelial Neoplasia, and for Prediction of Recurrence of Cervical Disease
Brief Title: Use of Human Papillomavirus Persistence for Determination of Treatment Efficacy Among Women With Cervical Dysplasia
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Swedish Cancer Society (Other)
Responsible Party: Anna Söderlund Strand, Dept. Medical microbiology, Malmö university hospital, 20502 Malmö, Sweden
Other Study IDs: 95-240
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Human Papillomavirus Infection; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical smear samples in physiologic saline.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives are to evaluate the effectiveness of treatment of cervical intraepithelial neoplasia (CIN) by loop electrosurgical excision procedure using persistence of human papillomavirus (HPV) as outcome, and to perform a long-term follow-up on the ability of HPV testing, as compared to cytology, to predict recurrence of high-grade CIN.

DETAILED DESCRIPTION:
Cervical samples for human papillomavirus (HPV) DNA analysis and cytological analysis were obtained from women with abnormal smears referred to Umeå university hospital, Sweden, for treatment with conization. These women were scheduled for HPV DNA testing and Pap smears before and 3, 6, 12, 24 and 36 months after treatment. The HPV DNA testing was performed with a PCR-based genotyping method.

ELIGIBILITY:
Inclusion Criteria:

* Referral to Umeå university hospital for treatment due to abnormal Pap smear.

Exclusion Criteria:

* Lack of informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 195 women referred for treatment of cervical intraepithelial neoplasia in the cathment area of Umeå university hospital. All women had abnormal smears at enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2001-02; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Söderlund Strand, PhD, Principal Investigator — Dept. medical microbiology, Malmö university hospital, Malmö, Sweden
Locations (1):
- Dept. obstetrics and gynecology, University hospital of Northern Sweden, Umeå, Sweden